CLINICAL TRIAL: NCT00179933
Title: The Impact of Implementing the Newborn Individualized Developmental Care and Assessment Program on Neurobehavioral Organization of Preterm Infants in the NICU
Brief Title: The Impact of Implementing NIDCAP on Preterm Infants in the NICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to fulfill intention of study, lost investigators.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Barbara Fleming, Clinical Nurse Specialist/Educator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-12574
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Infant, Premature
Keywords: developmental care; Neonatal Intensive Care Unit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Newborn Individualized Assessment Program

SUMMARY:
The purpose of this study is to evaluate the impact of the NIDCAP program of individualized patient consultation on the neurobehavioral organization of transported preterm infants in the NICU. Behavioral response to routine caregiving will be compared between infants in the pre-NIDCAP group to infants in the post-NIDCAP group. And it is this behavioral response that will be used to evaluate the effectiveness of the NIDCAP program.

DETAILED DESCRIPTION:
Therapies that have brought about sharp decreases in neonatal mortality have not brought about similar decreases in neurodevelopmental morbidity for preterm infants. Developmentally supportive care is NICU care that seeks to optimize the developmental course and outcomes for preterm infants. While other staff training programs for developmentally supportive care exist, it is the Newborn Developmental Care and Assessment Program (NIDCAP) that has been the methodology used in randomly controlled trials that demonstrate positive medical and neurobehavioral outcomes for preterm infants receiving developmentally supportive care. NICUs that care for all out-born or transported infants face unique challenges in balancing developmentally supportive nursing care with the high-technological medical needs of the most critically ill and extremely premature infants. Yet it is these most fragile infants who can most benefit from the positive impact the NIDCAP program can offer. Yet, there are no published studies documenting the impact of the NIDCAP program on neurobehavioral outcomes of these transported preterm infants exclusively.

Objectives: The objective of this project is to study the impact of implementing the NIDCAP program of individualized patient consultation on the neurobehavioral organization of transported preterm infants in the NICU of a major pediatric medical center.

Research Methods: A random sample of approximately 40 preterm infants will be recruited to participate in this descriptive study. In this phase-lag design, 20 infants will participate in the pre-NIDCAP intervention phase and 20 infants will participate in the post-NIDCAP intervention phase. Each infant within each phase will be videotaped during 2 routine nurse-caregiving sessions. The first session will occur within 72 hours of admission to the NICU at Children's Memorial Hospital (CMH). The second session will occur when the infant is 34-36 weeks corrected gestational age. The videotapes will be collected so that observations of the infant's physical environment and caregiving and an assessment of the infant's behavioral function can be scored randomly at the end of the study by an outside consultant without bias as to what phase the infant participated. In addition, demographic data will be collected on the sample infants. Data will be subjected to descriptive statistics, inferential statistics and correlational procedures.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born at less than or equal to 32 weeks gestation, appropriate for gestational age in weight

Exclusion Criteria:

* congenital or chromosomal abnormality, history of maternal substance abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Behavioral function score within 72 hours of admission and Behavioral function score at 34-36 weeks gestation.

SECONDARY OUTCOMES:
Environment and caregiving score within 72 hours of admit
Environment and caregiving score at 34-36 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Fleming, RNC, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Neonatal Intensive Care Unit Children's Memorial Hospital, Chicago, Illinois, United States